CLINICAL TRIAL: NCT04101890
Title: The Healthy Baby Bottoms Study: A Trial of Theraworx Foam Formulation for the Prevention and Treatment of Diaper Dermatitis
Brief Title: The Healthy Baby Bottoms Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator left the Institution and decision was made by funders to terminate the trial.
Sponsor: Linda Fu (Other)
Collaborators: Avadim Technologies, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Linda Fu, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 12239
Record Dates: First submitted 2019-09-16; First posted 2019-09-24 (Actual); Results first posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Diaper Dermatitis
MeSH Terms: conditions — Diaper Rash | interventions — Zinc Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaper care with Theraworx (Experimental): Participants will be given a 4 week supply of Theraworx Spray Foam, an FDA-registered OTC drug (NDC 61594-000), to apply a thin layer to their infant's entire diaper area with every diaper change (2-4 foam pumps or 4-6 sprays depending on the infant's size) for 4 weeks.
  Interventions: Drug: Diaper care with Theraworx
- Routine diaper care (No Intervention): Participants continue their typical diaper care.

INTERVENTIONS:
Drug: Diaper care with Theraworx — Theraworx foam formulation to be used as a preventive and treatment agent for diaper rashes
  Arms: Diaper care with Theraworx

SUMMARY:
Diaper dermatitis is one of the most common dermatologic diseases affecting infants and children. The incidence is highest among those 9-12 months old and it has been reported to affect 7-50% of infants in the US. It is caused by skin exposure to a combination of several factors including: excessive moisture, topical irritants, reduced pH, friction, maceration and bacterial infection. When infants soil their diaper, diaper contents saturate the area raising the pH of the skin above the normal level of 5 or less, and leaving the area highly vulnerable to maceration from friction. Irritants in urine and feces are then able to penetrate the macerated skin, causing inflammation and greater skin friability. An elevation in the skin pH allows pathogenic bacteria to overgrow, and combined with the breakdown in the skin's outer epithelial barrier, can lead to bacterial infection. Theraworx Foam Formulation-Allantoin Liquid by Avadim Technologies, Inc. is a skin protectant with use for temporary protection of minor cuts, scrapes, burns and chapped or cracked skin. As such, Theraworx Foam used in the diaper area may be beneficial for protecting skin against diaper rash wounds, as well as for assisting with wound healing and reducing any associated pain. The purpose of this study is to determine caregivers' perceptions of the benefits of using Theraworx Foam on their infant's diaper area as part of their hygienic routine, including whether they feel the product is pleasant and easy to use, and whether they feel it helps prevent and reduce the severity of diaper dermatitis in their infants 1-14 months old.

ELIGIBILITY:
Inclusion Criteria:

* Read English at the 8th grade level
* Have reliable access to email for 7 weeks
* Complete the first online survey within 24 hours of the request
* Custodial guardian of an infant between the ages of 1-12 months old living with him/her, wearing diapers, and has had ≥1 diaper rash in the 2 months preceding recruitment

Exclusion Criteria:

* Does not have a stable address at which to receive a package of Theraworx and is unable/unwilling to pick it up at Children's National Health System
* Infant is immunocompromised, has a congenital disorder, or on the day of recruitment, has a diaper rash, has a moderate to severe illness requiring hospitalization or transfer to the emergency room, or was circumcised <10 days prior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-01-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chidlren's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants completed routine diaper care during the run-in period, followed by diaper care with Theraworx during the experimental period.
Groups:
- Routine Diaper Care Followed by Diaper Care With Theraworx: Participants continue their typical diaper care for a period of 4 weeks. This is directly followed by 4 weeks of Theraworx Spray Foam, an FDA-registered OTC drug (NDC 61594-000), to apply a thin layer to their infant's entire diaper area with every diaper change (2-4 foam pumps or 4-6 sprays depending on the infant's size).
Period: Routine Diaper Care
Arm/Group | Routine Diaper Care Followed by Diaper Care With Theraworx
Started | 5
Completed | 5
Not Completed | 0
Period: Diaper Care With Theraworx
Arm/Group | Routine Diaper Care Followed by Diaper Care With Theraworx
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Routine Diaper Care Followed by Diaper Care With Theraworx: Participants continue their typical diaper care for 4 weeks followed immediately by 4 weeks of using Theraworx Spray Foam, an FDA-registered OTC drug (NDC 61594-000). During this second period, particpants apply a thin layer to their infant's entire diaper area with every diaper change (2-4 foam pumps or 4-6 sprays depending on the infant's size) for 4 weeks.
  Diaper care with Theraworx: Theraworx foam formulation to be used as a preventive and treatment agent for diaper rashes
Arm/Group | Routine Diaper Care Followed by Diaper Care With Theraworx
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: months] | 7 [5 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Frequency of diaper rash in last 30 days, continuous [Median (Inter-Quartile Range); unit: days] | 7 [5 to 20]

OUTCOME MEASURES:

1. Primary Outcome: Caregiver's Self-report of Prevention of Diaper Dermatitis in Infant
Description: Caregivers self-report on a weekly basis the total number of days during the past week that their infant had a diaper rash. Diaper rash was defined as the presence of one or more of the following in the diaper region: redness, skin breakdown, papules or pustules. The total number of days with diaper rash for the entire 4 week period was summed from the 4 weekly surveys (outcome measure range: 0-28 days with fewer days representing a better outcome).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: days
Groups:
- Routine Diaper Care Followed by Diaper Care With Theraworx: Participants continue their typical diaper care x4 weeks, immediately followed by a 4 week period of using Theraworx Spray Foam, an FDA-registered OTC drug (NDC 61594-000). During this second period, particpants apply a thin layer to their infant's entire diaper area with every diaper change (2-4 foam pumps or 4-6 sprays depending on the infant's size) for 4 weeks.
Arm/Group | Routine Diaper Care Followed by Diaper Care With Theraworx
Number analyzed (Participants) | 5
days
  Routine Diaper Care | 3.7 (2.5)
  Diaper care with Theraworx | 1.7 (1.5)

2. Secondary Outcome: Caregiver's Self-report of Diaper Rash Severity
Description: Caregivers used a modified Diaper Dermatitis Scale (Buckley, et al, Pediatric Dermatology 2016) to report infant diaper rash severity. The scale ranged from 0 (none) to 6 (most severe) with higher scores indicating a worse outcome. Items on the scale included assessments of rash size (0-2), redness (0-1), evidence of skin breakdown (0-1), evidence of papules (0-1) and evidence of pustules (0-1). Mean score was calculated using scores for every day over 28 days.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Routine Diaper Care Followed by Diaper Care With Theraworx: Participants continued their typical diaper care for 4 weeks immediately followed by 4 weeks of using Theraworx Spray Foam, an FDA-registered OTC drug (NDC 61594-000). During the second period, participants applied a thin layer to their infant's entire diaper area with every diaper change (2-4 foam pumps or 4-6 sprays depending on the infant's size).
Arm/Group | Routine Diaper Care Followed by Diaper Care With Theraworx
Number analyzed (Participants) | 5
score on a scale
  Routine Diaper Care | 4.45 (3.35)
  Diaper Care with Theraworx | 3.15 (3.82)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Diaper Care With Theraworx | Routine Diaper Care
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT04101890/Prot_SAP_000.pdf